CLINICAL TRIAL: NCT00995098
Title: The Impact of Early Enteral Nutrition on the Clinical Outcomes of Severe Acute Pancreatitis Patients: A Randomized Control Trial
Brief Title: Early Enteral Nutrition for Severe Acute Pancreatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sichuan Academy of Medical Sciences (Other)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Bin Cai/Deputy Chief, Sichuan Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAMS-080384
Record Dates: First submitted 2009-10-11; First posted 2009-10-15 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Acute Necrotizing Pancreatitis
Keywords: Acute severe pancreatitis; nutritional support; enteral nutrition; parenteral nutrition
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing; Hyperphagia | interventions — Parenteral Nutrition; NovaMin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early enteral nutrition (Experimental): Twenty patient will be enrolled into this arm. Enteral nutrition administration will start within 24 hours after admission through naso-jejunal tube and continue for 7 days after admission.Naso-jejunal tube will be set up by endoscopy.
  Interventions: Dietary Supplement: early enteral nutrition
- Control: Parenteral Nutrition (Active Comparator): Twenty patient will be enrolled into this arm. PN administration will start within 24 hours after admission and continue for 7 days after admission.Parenteral nutrition will be administered through subclavian central venous catheter.
  Interventions: Dietary Supplement: Parenteral nutrition

INTERVENTIONS:
Dietary Supplement: early enteral nutrition — Enteral nutrition will be administered within 24 hours of admission through naso-jejunal tube and continue for 7 days after admission. Naso-jejunal tube will be set up by endoscopy. X-ray will be used to place the distal end of the feeding tube and EN would not start until the distal end of the feeding tube has been placed at the remote end of Treitz ligament. Standard enteral nutrition liquid regimen (Nutrison Fibre) will be used. Patients are targeted to receive calories for 25 kcal/kg/day and nitrogen for 0.2g/kg/day.
  Other Names: Nutrison Fibre
  Arms: Early enteral nutrition
Dietary Supplement: Parenteral nutrition — PN administration will start within 12 hours of admission and continue for 7 days after admission. Patients will receive calories for 25 kcal/kg and nitrogen for 0.2g/kg. Twenty percent of the calories will be provided by fat emulsion (LCT/MCT) and the remaining will be provided by dextrose. Nitrogen will be provided by balanced amino acids injection (Novamin). All PN components will be compounded into 3-liters bags under sterile conditions. Nutrition regimen will be administered through subclavian central venous catheter.
  Other Names: Lipovenoes(LCT/MCT fat emulsion, 20%); Novamin (11.4%)
  Arms: Control: Parenteral Nutrition

SUMMARY:
There is increasing evidence that indicates early enteral nutrition may be associated with improved outcome in acute pancreatitis patients. However, most of the clinical trials regarding this targeted mild to moderated pancreatitis patients. In regard to severe acute pancreatitis (SAP) patients, current results from randomized control trials (RCTs) are inconclusive. The researchers of this study aim to investigate the impact of early enteral nutrition on the clinical outcomes of SAP patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of severe acute pancreatitis
* Consent informed

Exclusion Criteria:

* Diabetes mellitus
* Allergy for any ingredient of PN or EN regimen
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
All cause mortality | Three months

SECONDARY OUTCOMES:
Pancreatic sepsis | Three months
Length of hospitalization | From admission to discharge
Operation ratio | From admission to discharge
Cost of hospitalization | From admission to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Bin Cai, M.D, Study Director — Sichuan Academy of Medical Sciences; Hua Jiang, M.D, Principal Investigator — Sichuan Academy of Medical Sciences; Jun Zeng, M.D, Study Chair — Sichuan Academy of Medical Sciences
Locations (1):
- Sichuan Academy of Medical Sciences, Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

REFERENCES:
- [Background] Marik PE, Zaloga GP. Meta-analysis of parenteral nutrition versus enteral nutrition in patients with acute pancreatitis. BMJ. 2004 Jun 12;328(7453):1407. doi: 10.1136/bmj.38118.593900.55. Epub 2004 Jun 2. PMID 15175229
- [Background] Meier R, Beglinger C, Layer P, Gullo L, Keim V, Laugier R, Friess H, Schweitzer M, Macfie J; ESPEN Consensus Group. ESPEN guidelines on nutrition in acute pancreatitis. European Society of Parenteral and Enteral Nutrition. Clin Nutr. 2002 Apr;21(2):173-83. doi: 10.1054/clnu.2002.0543. No abstract available. PMID 12056792
- [Background] McClave SA, Chang WK, Dhaliwal R, Heyland DK. Nutrition support in acute pancreatitis: a systematic review of the literature. JPEN J Parenter Enteral Nutr. 2006 Mar-Apr;30(2):143-56. doi: 10.1177/0148607106030002143. PMID 16517959